CLINICAL TRIAL: NCT05816993
Title: Assessment of Neurological Manifestations in Gaucher Disease Patients Attending Assiut University Children's Hospital
Brief Title: Assessment of Neurological Manifestations in Gaucher Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gehan Mohamed Galal, Principle investigatir, Assiut University
Other Study IDs: Neurological signs in Gaucher
Record Dates: First submitted 2023-03-30; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current work aims to detect the frequency and types of neurological disorders in patient diagnosed as Gaucher disease in Assiut University Children's Hospital

DETAILED DESCRIPTION:
Gaucher disease, the most common lysosomal storage disorder, caused by reduced activity of acid β-glucosidase and mutations in the GBA1 gene. This leads to the accumulation of its normal substrate, glucocerebroside, in tissue macrophages, affecting the hematological, visceral, bone and neurologic systems. The determination of deficient β-glucocerebrosidase activity in leukocytes or fibroblasts by enzymatic assay is the gold standard for the diagnosis of Gaucher disease. Clinically, Gaucher disease is classified into three major forms based upon the absence or presence and rate of progression of neurological manifestations : type 1 (non-neuronopathic), type 2 (acute neuronopathic), and type 3 (subacute neuronopathic). The nGD forms are Gaucher disease type 2 (GD2) and Gaucher disease type 3 (GD3). GD2 is the acute neuronopathic form and has an early onset CNS involvement, typically manifesting in the first 6 months of life and leading to death by age 2 years, although patients may live up to age 4 years or beyond with supportive medical care. GD3, or the chronic neuronopathic form, has a slightly later onset, CNS symptoms typically manifesting months to years after birth, and has a much slower neurological progression than is seen in GD2. GD3 is the predominant form of Gaucher disease. Phenotypically, there is a wide spectrum of visceral and neurological manifestations. Enzyme replacement therapy has been shown to be effective in reducing glucocerebroside storage burden and diminishing the deleterious effects caused by its accumulation. Enzyme replacement is effective in managing the visceral disease; however, treating the neurological manifestations has proved to be more challenging. Currently, there is no agreement on a definition of nGD, other than one by exclusion ("the presence of neurological involvement in a patient with biochemically proven Gaucher disease, for which there is no explanation other than Gaucher disease")

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Gaucher Disease

Exclusion Criteria:

* Not meeting Inclusion criteria

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Gaucher disease patients from age 1m to age 18y with neurological manifestations
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with neurological disorders in pediatric patients diagnosed as Gaucher disease | Baseline
  Types of neurological disorders in patients with Gaucher disease

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ghazaly, Prof, Principal Investigator — Assiut University; Mostafa Embaby, Prof, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No